CLINICAL TRIAL: NCT06994130
Title: A Prospective Evaluation of Seravue Device Sensitivity and Specificity for Surveillance and Diagnosis of Patients at Risk for Hepatocellular Carinoma (HCC)
Brief Title: Seravue Validation Study for Hepatocellular Carcinoma (HCC) Diagnosis
Acronym: Seravue
Status: Not yet recruiting | Type: Observational
Sponsor: ImCare Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: IMC001
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Hepatic Cancer
Keywords: liver cancer; AFP; ultrasound
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Group 1: Patient under surveillance for hepatocellular carcinoma coming in every 6 months for an ultrasound and AFP
  Interventions: Diagnostic Test: Seravue

INTERVENTIONS:
Diagnostic Test: Seravue — . This study seeks to test the performance of the SeravueTM (LC-SPIK) device alone or in combination with ultrasound as a tool for HCC surveillance in diverse patient populations and clinical settings.

SUMMARY:
Currently, ultrasound with or without AFP is the standard of care when it comes to surveillance for HCC in high-risk populations. While ultrasound is non-invasive and plays a critical role in detecting HCC, it is operator-dependent, inconvenient, and may have access issues in low-resource settings. Most critically, ultrasound is not sensitive enough to detect or confirm HCC in its most critical early stages, where treatment options are most effective and result in the best patient outcomes. AFP on the other hand, suffers from poor sensitivity and specificity generally, and its performance is insufficient for use as a surveillance tool. There remains a clear unmet need for a blood test that is sensitive enough to detect HCC in its early stages while being cost-effective and accessible for use as a surveillance tool.

The investigators have previously demonstrated that serum liver cancer-secreted serine protease inhibitor Kazal (LC-SPIK) can reliably detect early HCC in addition to differentiating between it and other liver diseases. This study seeks to test the performance of the Seravue (LC-SPIK) device alone or in combination with other HCC diagnostic tests as a tool for HCC surveillance in diverse patient populations and clinical settings.

DETAILED DESCRIPTION:
Patients who meet eligibility criteria and provide written informed consent will undergo comprehensive screening evaluations and standard of care clinical laboratory tests, including hepatic ultrasound and AFP testing at baseline, 6, 12, and 18 months after enrollment, or until the diagnosis of HCC. At each visit, blood specimens will be collected for testing with the Seravue device and for clinical and study biomarker testing including AFP. Pateints negative for ultrasound, AFP or Seravue results will continue on with the study. Patient testing positive for ultrasound, or AFP test results will undergo CT [with or without contrast] or MRI imaging to determine the presence or absence of HCC. Inconclusive or indeterminate radiographic diagnosis of HCC will require repeated imaging or lesion biopsy and histopathologic diagnosis to confirm or exclude the presence of HCC per standard of care guidelines. Once HCC diagnosis is confirmed, the patient will exit the study. A patient that demonstrates positive test for Seravue will return to the study visit schedule with no action being taken. All patients will have their medical records reported at month 24 for any new cancer diagnosis and standard of care labs performed. Adverse events (AEs) and serious adverse events (SAEs) will not be collected.

ELIGIBILITY:
INCLUSION/EXCLUSION CRITERIA:

Patients who provide written informed consent and meet eligibility criteria will undergo baseline assessments and be entered into the study.

Inclusion Criteria:

A patient must meet all of the following criteria to be eligible for this study:

1. The patient is willing and able to provide signed informed consent.
2. The patient is aged ≥21to ≤84 years.
3. The patient is willing to undergo phlebotomy and provide blood samples for future biomarker analysis.
4. The patient is willing and able to undergo regularly scheduled onsite liver cancer surveillance by ultrasound and AFP and any resulting axial imaging such as computed tomography (CT, with or without contrast), magnetic resonance imaging (MRI), or ultrasound per the standard of care guidelines and study protocol schedule.
5. The patient has been diagnosed with hepatic cirrhosis of any etiology (both viral and non-viral), or Hepatitis B Virus (HBV). This includes HBV patients with pre-existing cirrhosis prior to antiviral therapy or other treatments leading to fibrosis regression who continue to be at risk.

   a. Cirrhosis may be diagnosed by any one of the following three methods: i. Biopsy and histological examination ii. Fibroscan (VCTE ≥ 12.5kPa) for all etiologies except HBV), Magnetic resonance elastography (≥ 4 kPa) iii. A combination of imaging (MRI, CT, or ultrasound) demonstrating a cirrhotic appearing liver AND at least one of the following:

1. Thrombocytopenia 2. Clinical symptoms (including but not limited to ascites, portal hypertension, hypersplenism, esophageal varices, and encephalopathy).

6) The patient has been diagnosed with HBV without cirrhosis.

1. HBV will be defined by either a positive blood test for HBsAg, quantitative HBsAg, HBeAg OR detectable HBV DNA prior to initiating antiviral therapy.
2. Patients are:

i. Asian males ≥ 40 years old OR ii. Asian females ≥ 50 years old OR iii. Patients of any ethnicity with a page B score ≥ 10

Exclusion Criteria

A patient who meets any of the following criteria will be excluded from this study:

1. Any health condition or other reason which, in the opinion of the investigator, would prelude study participation.
2. Current Child Pugh C cirrhosis
3. The patient has previously been diagnosed with a primary liver cancer or any cancer that has metastasized.
4. The patient has participated in an interventional clinical study within 30 days prior to screening in which an experimental treatment was administered.
5. The patient is unable or unwilling to submit to phlebotomy for testing or undergo ultrasound or other diagnostic imaging such as contrast-enhanced CT or MRI as recommended by AASLD standard of care guidelines.
6. The patient would not routinely be recommended for HCC surveillance.
7. The female patient is pregnant or plans to become pregnant during the study.
8. History of solid nodule on baseline ultrasound (i.e., lesion 1cm or greater) within 9 months prior to consent without subsequent diagnostic multi-phase CT/MRI demonstrating benign nature
9. AFP >20 ng/mL within 6 months prior to consent, in the absence of a contrast-enhanced multi-phase CT or MRI (before or after) in the past year demonstrating lack of suspicious liver lesions.

   a. If the AFP is >20 ng/mL during the study, the patient should undergo a contrast-enhanced multi-phase CT or MRI. if the patient has consistent elevations that are not increasing, repeat diagnostic testing will be left to the discretion of the investigator or the faculty.
10. History of LR-4, LR-5, or LR-M on multi-phase CT or contrast-enhanced MRI prior to consent
11. Patient's provider is planning to use only MRI- or CT- based surveillance moving forward
12. History of Fontan associated liver disease or cardiac cirrhosis
13. Actively listed for liver transplantation

Ages: 21 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient under surveillance for HCC
Sampling Method: Probability Sample
Enrollment: 1392 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | From enrollment to the end of study 24 months
  The primary objective of the study is to test that the sensitivity of the SeravueTM test in conjunction with ultrasound (LC-SPIK+US) is higher compared to a point-estimate of the sensitivity of the standard of care (US+AFP) in detecting HCC for patients with high risk of HCC due to chronic HBV or hepatic cirrhosis while the specificity are similar

SECONDARY OUTCOMES:
Secondary Objective | From enrollment to the end of study 24 months
  * • To test that the sensitivity of the SeravueTM test alone is higher compared to a point estimate of the sensitivity of the ultrasound alone in detecting HCC for patients with high risk of HCC due to chronic HBV or hepatic cirrhosis, while the specificity is similar.
  * To test that the sensitivity of the SeravueTM test alone is higher compared to a point estimate of the sensitivity of the standard of care (US+AFP) in detecting HCC for patients with high risk of HCC due to chronic HBV or hepatic cirrhosis

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No